CLINICAL TRIAL: NCT02999581
Title: Effects of a Pre-Workout Dietary Supplement on Training Adaptations in Resistance Trained Athletes
Brief Title: Effects of a Pre-Workout Dietary Supplement on Training Adaptations
Acronym: NB2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Nutrabolt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2014-0079FX
Record Dates: First submitted 2016-12-16; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Dietary Modification

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- C4 Extreme (Experimental): One dose of 12 grams (powder mixed with water): 1500 mg beta alanine, 1000 mg creatine nitrate, 1000 mg arginine alpha-ketoglutarate, 250 mg vitamin C, 150 mg N-Acetyl-Tyrosine, 135 mg caffeine, 7.5 mg L-Dopa, 30 mg vitamin B3, 10 mg Bitter Orange (Citrus Aurantium) fruit standardized for 30% synephrine (Advantra Z), 0.5 mg vitamin B6, 0.25 mg vitamin B9, and 0.035 mg vitamin B12.
  Interventions: Dietary Supplement: C4 Extreme, C4 Extreme (without Advantra Z)
- C4 Extreme (without Advantra Z) (Active Comparator): One dose of 12 grams (powder mixed with water): 1500 mg beta alanine, 1000 mg creatine nitrate, 1000 mg arginine alpha-ketoglutarate, 250 mg vitamin C, 150 mg N-Acetyl-Tyrosine, 135 mg caffeine, 7.5 mg L-Dopa, 30 mg vitamin B3, 0.5 mg vitamin B6, 0.25 mg vitamin B9, and 0.035 mg vitamin B12.
  Interventions: Dietary Supplement: C4 Extreme, C4 Extreme (without Advantra Z)
- Placebo (Placebo Comparator): One dose of flavored placebo (powder mixed with water)
  Interventions: Dietary Supplement: C4 Extreme, C4 Extreme (without Advantra Z)

INTERVENTIONS:
Dietary Supplement: C4 Extreme, C4 Extreme (without Advantra Z)

SUMMARY:
The purpose of this study is to examine the effects of a pre-workout dietary supplement during resistance training on training adaptations.

DETAILED DESCRIPTION:
A number of nutritional strategies have been developed to optimize nutrient delivery prior to exercise. This includes providing carbohydrate and a number of ergogenic nutrients prior to, during and/or following exercise. As a result, a number of pre-workout supplements have been developed to increase energy availability, promote vasodilation and/or positively affect exercise capacity. The purpose of this study is to investigate the effects of ingesting a pre-workout dietary supplement during resistance training on training adaptations.

ELIGIBILITY:
Inclusion Criteria:

* you are an apparently healthy and recreationally active male between the ages of 18 and 40.
* you will need to have at least six months immediate prior history of resistance training on the bench press and leg press or squat.

Exclusion Criteria:

* you have a history of treatment for metabolic disease (i.e., diabetes), hypertension, hypotension, thyroid disease, arrhythmia and/or cardiovascular disease;
* you are currently using prescription medications;
* you have an intolerance to caffeine and/or other natural stimulants;
* you have a history of smoking;
* you drink excessively (i.e., 12 drinks per week or more);

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Examine the effects of C4 supplementation during resistance training by assessing body water | Eight weeks
Examine the effects of C4 supplementation during resistance training by assessing body composition | Eight weeks
Examine the effects of C4 supplementation during resistance training by assessing macronutrient intake | Eight weeks
Examine the effects of C4 supplementation during resistance training by assessing 1 RM (repetition maximum) strength | Eight weeks
Examine the effects of C4 supplementation during resistance training by assessing anaerobic sprint capacity | Eight weeks
Examine the effects of C4 supplementation during resistance training by assessing muscle creatine levels | Eight weeks
Examine the effects of C4 supplementation during resistance training by assessing muscle carnosine levels | Eight weeks
Examine the effects of C4 supplementation during resistance training by assessing cognitive function (i.e., Stroop Color and Word Test, Word Recall Test and Readiness to perform VAS) | Eight weeks

SECONDARY OUTCOMES:
Measure standard clinical chemistry panels in the blood to evaluate safety | Eight weeks
Record side effects to evaluate safety | Eight weeks
Measure heart rate to evaluate safety | Eight weeks
Measure blood pressure to evaluate safety | Eight weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung YP, Earnest CP, Koozehchian M, Cho M, Barringer N, Walker D, Rasmussen C, Greenwood M, Murano PS, Kreider RB. Effects of ingesting a pre-workout dietary supplement with and without synephrine for 8 weeks on training adaptations in resistance-trained males. J Int Soc Sports Nutr. 2017 Jan 3;14:1. doi: 10.1186/s12970-016-0158-3. eCollection 2017. PMID 28096757